CLINICAL TRIAL: NCT00534534
Title: Randomized Clinical Trial of the Effect of Standard Versus Intensive Intervention Protocol in Attempting to Reduce Recurrent Episodes of Acute Alcoholic Pancreatitis
Brief Title: Decrease of Recurrent Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R00126A
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Pancreatitis
Keywords: Pancreatitis; acute; alcoholic; recurrence; alcoholism; treatment; Acute alcoholic pancreatitis
MeSH Terms: conditions — Pancreatitis; Recurrence; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): All these patients will be advised, i.e. undergo behavioural intervention, against alcohol use in the standard fashion. No drugs will be used. In addition, they also will undergo repeated similar interventions at 6 mo intervals. They are re-examined at two years for alcohol consumption and for the number of recurrent pancreatitis during the two year period.
  Interventions: Behavioral: Repeated behavioural intervention without any drugs
- Standard (No Intervention): All these patients will be advised, i.e. undergo behavioural intervention, against alcohol use in the standard fashion. No drugs will be used. They are re-examined at two years for alcohol consumption and for the number of recurrent pancreatitis during the two year period.

INTERVENTIONS:
Behavioral: Repeated behavioural intervention without any drugs — All these patients will be advised, i.e. undergo "behavioural intervention", against alcohol use in the standard fashion as those in the standard group. No drugs will be used as part of the intervention. They also will undergo repeated interventions at outpatient visits at 6 mo intervals. They are re-examined at two years for alcohol consumption and for the number of recurrent pancreatitis during the two year period.
  Arms: 1

SUMMARY:
Retrospective studies have shown, that about half of the patients will have a recurrent episode after the first acute alcoholic pancreatitis. Of the patients in hospital, more than half annually are treated for recurrent acute pancreatitis. Because alcohol has been shown an important factor in the development of recurrent pancreatitis, it was hypothesized, that by attempting intensively to diminish the individual alcohol consumption the number of recurrent pancreatitis could be decreased. Two protocols will be compared: A) initial intervention against alcohol abuse and B) repeated interventions at 6 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recovered from their first acute alcoholic pancreatitis and start to be ready to be discharged from hospital

Exclusion Criteria:

* Other etiologies of pancreatitis besides alcohol
* Uncertain diagnosis
* Recurrent disease
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2001-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The number of recurrent pancreatitis during the study period | 2 years

SECONDARY OUTCOMES:
Decrease of alcohol consumption | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isto H Nordback, M.D., Study Chair — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland